CLINICAL TRIAL: NCT07008053
Title: BR (Bendamustine and Zuberitamab) Combined With OR (Orelabrutinib and Zuberitamab) in Treatment-naïve Marginal Zone Lymphoma: A Multicenter, Prospective Study
Brief Title: BR Combined With OR in Treatment-naïve Marginal Zone Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BROAD
Record Dates: First submitted 2025-05-18; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Marginal Zone Lymphomas
Keywords: Lymphoma、Marginal zone lymphoma、Orelabrutinib; Bendamustine; Zuberitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BR (bendamustine and zuberitamab) + OR (orelabrutinib and zuberitamab) (Experimental): Induction therapy: patients will receive 90 mg/m2 of bendamustine and 375 mg/m2 zuberitamab from cycles 1 to 3, followed by 150 mg of orelabrutinib and 375 mg/m2 zuberitamab from cycles 4 to 6.
  Maintenance therapy: at the investigator's discretion, patients who achieved a complete response or partial response could be assigned to maintenance therapy, consisting of 150 mg of orelabrutinib for 24 cycles.
  Interventions: Drug: BR+OR

INTERVENTIONS:
Drug: BR+OR — Patients who meet the inclusion criteria will enter the treatment period, which consists of an induction phase followed by a maintenance phase. During the induction treatment period, a combined treatment of 3 cycles of the BR regimen and 3 cycles of the OR regimen will be administered, every 28-day cycle for 6 cycles. After the induction treatment, the efficacy assessment will determine whether patients with CR or PR proceed to the maintenance treatment period. Orelabrutinib monotherapy will used as maintenance therapy, every 28-day cycle for up to 24 cycles, or until disease progression/recurrence, unacceptable toxicity, death or consent withdrawal.

SUMMARY:
This is a multi-center, prospective study. The main purpose is to evaluate the efficacy and safety of BR (bendamustine and zuberitamab) combined with OR (orelabrutinib and zuberitamab) in treatment-naïve patients with marginal zone lymphoma.

DETAILED DESCRIPTION:
Marginal zone lymphoma (MZL) represents the second most prevalent indolent lymphoma subtype, accounting for 5-15% of all non-Hodgkin lymphomas. MZL is categorized into three subtypes based on distinct clinical and pathological features: mucosa-associated lymphoid tissue lymphoma (MALT), nodal marginal zone lymphoma (NMZL), and splenic marginal zone lymphoma (SMZL). Currently, there remains no internationally recognized consensus regarding the optimal first-line treatment for MZL. Exploring more effective, low-toxicity treatment regimens for MZL patients is a scientifically valuable and clinically significant attempt. Orelabrutinib, a novel highly selective BTK inhibitor, has been approved by the NMPA for the treatment of MZL in patients who have received at least one prior treatment.

This study is a multi-center, prospective clinical study involving previously untreated MZL patients. During the induction therapy phase, patients will receive 90 mg/m2 of bendamustine and 375 mg/m2 zuberitamab from cycles 1 to 3, followed by 150 mg of orelabrutinib and 375 mg/m2 zuberitamab from cycles 4 to 6. At the investigator's discretion, patients who achieved a complete response or partial response could be assigned to maintenance therapy, consisting of 150 mg of orelabrutinib for up to 24 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, gender not limited;
2. Histopathologically confirmed CD20-positive marginal zone lymphoma including MALT, SMZL, NMZL;
3. At least one measurable lesion;
4. Ann Arbor stage II includes abdominal or intestinal tumor invasion, stage III and IV have indications for treatment (e.g. B symptoms, decreased blood cells, bleeding, large masses, rapid tumor progression);
5. Without systemic treatment, MZL that has progressed, recurred, or is not suitable for local treatment after previous local treatment (local treatments include surgery, radiotherapy, Helicobacter pylori treatment, hepatitis C treatment, and CD20 monoclonal antibody monotherapy);
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
7. Major organ function meets the following criteria: a) Complete blood count: Absolute neutrophil count ≥1.5×10^9/L, platelets ≥75×10^9/L, hemoglobin ≥75g/L; if accompanied by bone marrow invasion, absolute neutrophil count ≥1.0×10^9/L, platelets ≥50×10^9/L, hemoglobin ≥50g/L; b) Blood biochemistry: Total bilirubin ≤1.5 ULN, AST or ALT ≤2 ULN; serum creatinine ≤1.5 ULN;
8. Coagulation function: International normalized ratio (INR) ≤1.5 ULN;
9. Expected survival time ≥12 months;
10. Voluntarily sign a written informed consent form before the trial screening.

Exclusion Criteria:

1. Currently or previously diagnosed with other malignant tumors, unless curative treatment has been performed and there is evidence of no recurrence or metastasis within the last 5 years;
2. Lymphoma involving the central nervous system or transformation to a higher grade;
3. Have uncontrolled or significant cardiovascular disease: a) Within 6 months prior to the first dose of the study drug, there was New York Heart Association (NYHA) Class II or above congestive heart failure, unstable angina, myocardial infarction, or any arrhythmia requiring treatment at screening, with a left ventricular ejection fraction (LVEF)<50%; b) Primary cardiomyopathy (e.g., dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, or unclassified cardiomyopathy); c) History of clinically significant QTc interval prolongation, or QTc interval >470 ms for females and >450 ms for males during the screening period; d) Subjects with symptomatic or pharmacologically treated coronary artery disease; e) Subjects with uncontrolled hypertension (blood pressure not reaching target despite lifestyle modifications and the use of reasonable, tolerable doses of 3 or more antihypertensive drugs (including diuretics) for over 1 month, or blood pressure only effectively controlled with 4 or more antihypertensive drugs.
4. Active bleeding within 2 months prior to screening, or currently taking anticoagulant medications, or the investigator considers there to be a definite bleeding tendency;
5. History of deep vein thrombosis or pulmonary embolism within the past six months.
6. Major surgery within 6 weeks prior to screening or minor surgery within 2 weeks prior to screening. Major surgery is defined as any surgical procedure that requires general anesthesia, except endoscopic procedures performed for diagnostic purposes, which are not considered major surgery
7. Active infection or uncontrolled HBV (positive for HBsAg and/or HBcAb and positive for HBV DNA titer), HCV Ab positive, HIV/AIDS, or other serious infectious diseases;
8. Patients currently have pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonia, or other conditions affecting lung function；
9. Pregnant or lactating women and women of childbearing age who are unwilling to take contraceptive measures;
10. Need to continuously take drugs with moderate to severe inhibitory or strong inductive effects on cytochrome P450 CYP3A;
11. Other conditions that the investigator considers unsuitable for participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | From enrollment to the end of induction therapy of cycle 6 (each cycle is 28 days)
  Complete response rate is defined as the proportion of patients with a response of CR.

SECONDARY OUTCOMES:
Overall response rate (ORR) | At the end of induction therapy (6 cycles; each cycle is 28 days)
  The ORR is defined as the proportion of patients with a response of CR or PR.
Time to response (TTR) | From the start of therapy to the first documentation of response, assessed up to 3 years.
  TTR is defined as the time from the start of therapy to the first response.
Duration of Response (DOR) | From the first demonstration of response until disease progression/death, up to 3 years
  DOR is defined as the time from documentation of response to treatment to the first documentation of tumor progression or death due to any cause, whichever comes first.
Progression-free survival (PFS) | From the date of enrollment until the date of first documented progression, up to 3 years
  PFS is defined as the time from enrollment to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. PFS for patients without disease progression, relapse, or death will be censored at the time of the last tumor assessment.
Overall survival (OS) | From the date of enrollment until the date of death, up to 3 years
  OS is defined as the enrollment to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
The occurrence of adverse events (AEs) | From the date of enrollment until the date of death, up to 3 years
  AEs will be graded by the investigator according to the NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Huilai Zhang, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (6):
- China (6):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin